CLINICAL TRIAL: NCT02285192
Title: Positron Lymphography Via Intracervical 18F-FDG Injection for Pre-surgical Lymphatic Mapping in Stage IB1 Cervical Cancer and High-grade Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-222
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer; Endometrial Cancer
Keywords: 18F-FDG Injection; Positron Lymphography; Lymphatic Mapping; sentinel lymph nodes; PET/CT; 14-222
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Fluorodeoxyglucose F18

ARMS (1):
- intracervical 18F-FDG injection during a dynamic PET/CT (Experimental): The first 20 eligible patients will be consented to undergo intracervical 18F-FDG injection during a dynamic PET/CT scan. Study enrollment will occur in the clinic during the visit in which they are consented for surgery. Recruited patients will undergo 18F-FDG-guided PET imaging on the day of their scheduled staging surgery. The experimental PET/CT is anticipated to take 2 hours. The second stage of accrual will replace PET/CT with PET/MRI imaging. In every other aspect, patients will receive standard peri- and postoperative care.
  Interventions: Radiation: 18F-Fluorodeoxyglucose (18F-FDG); Device: PET/CT imaging; Device: PET/MRI imaging

INTERVENTIONS:
Radiation: 18F-Fluorodeoxyglucose (18F-FDG)
Device: PET/CT imaging
Device: PET/MRI imaging

SUMMARY:
The purpose of this study is to see if a radioactive substance called 18F-Fluorodeoxyglucose (18F- FDG), injected into the cervix during a PET/CT scan done before surgery can show us more clearly which lymph nodes in the pelvis (the area near your uterus and cervix) contain cancer.

ELIGIBILITY:
Inclusion Criteria:

* The study population will include women with stage IB1 cervical cancer (any histologic subtype) deemed eligible for surgery, and women with a clinical stage I high-grade endometrial cancer planning to undergo surgical staging. High grade is defined by the following:

  * Uterine serous carcinoma
  * Clear cell endometrial carcinoma
  * Grade 3 endometrioid carcinoma
  * Endometrial carcinosarcoma
  * Clinical stage I grade 1-2 endometrial cancer also eligible with deep myoinvasion ≥ 50% shown on preop MRI and/or elevated preop CA-125 > 35 U/ml.
* Age ≥18 years
* Hemoglobin ≥10 g/dL
* Plasma albumin ≥3 g/dL
* GOG performance status ≤2
* Plasma glucose ≤200 mg/dL
* Plasma creatinine ≤1.6
* Well-controlled hypertension
* Medical clearance for surgery and considered an appropriate surgical candidate
* Negative serum pregnancy test, if of child-bearing potential
* If, based on surgeon's assessment, the patient is recommended to undergo surgical staging for histologically confirmed endometrial cancer or if IB1 cervical cancer is deemed eligible for surgical treatment of disease
* Participation in other research protocols does not exclude a patient from participation in this study

Exclusion Criteria:

* Hemoglobin <10 g/dL
* Plasma albumin <3 g/dL
* GOG performance status >2
* Plasma glucose >200 mg/dL
* Renal insufficiency with plasma creatinine >1.6
* Uncontrolled hypertension
* Patient does not meet medical clearance for surgery and is not considered an appropriate surgical candidate
* Pregnancy

For Stage 2:

* Patient who are unwilling or unable to undergo MRI including patients with contraindications to MRI such as the presence of cardiac pacemakers of non-compatible intracranial vascular clips, claustrophobia, inability to lie flat for the duration of the study etc.
* Patients with a metallic hip implant or any other metallic implant or device in the pelvis that might distort local magnetic field and compromise quality of MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of Positron Lymphography | 2 years
  Accuracy of Positron Lymphography will be defined in terms of sensitivity and will consist of pathology review of labelled, excised specimens compared with lymph node imaging data acquired preoperatively.

SECONDARY OUTCOMES:
to evaluate several standard uptake value (SUV) (18F-FDG avidity) | 2 years
  will assess the ability of SUV to predict malignant disease. The continuous variable of SUV assigned to a given lymph node during Positron Lymphography will be compared with the pathologic assessment (benign vs malignant) of each labelled lymph node. The SUV assigned to a given lymph node is done using the the imaging software and not up to the discretion of the radiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mueller, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/